CLINICAL TRIAL: NCT01530139
Title: Personalised Nutrition: An Integrative Analysis of Opportunities and Challenges
Brief Title: Strategies for Personalised Nutrition
Acronym: Food4Me
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: University College Dublin (Other); Maastricht University (Other); University of Oslo (Other); University of Navarra (Other); Harokopio University (Other); University of Reading (Other); National Food and Nutrition InstitutE (Unknown); Technical University of Munich (Other); University of Newcastle Upon-Tyne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Food4Me-549426
Record Dates: First submitted 2012-02-01; First posted 2012-02-09 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Eating; Diet; Phenotype; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Level 0 (Placebo Comparator): Level 0: Control group - participants will receive non-personalized dietary advice for improved food choice based on standard population healthy eating guidelines.
  Interventions: Behavioral: Level 0
- Level 1 (Experimental): Level or Group 1: participants will receive personalised dietary advice based on their dietary intake data alone.
  Interventions: Behavioral: Level 1
- Level 2 (Experimental): Level or Group 2: participants will receive personalised dietary advice taking their dietary intake and phenotypic data ( obesity-related phenotypes and clinical biomarkers) into account.
  Interventions: Behavioral: Level 2
- Level 3 (Experimental): Level or Group 3 : participants will receive personalised dietary advice taking their dietary intake, phenotypic (obesity-related markers) and genotypic data into account.
  Interventions: Behavioral: Level 3

INTERVENTIONS:
Behavioral: Level 1 — Level 1 - Participants will receive personalised dietary advice based on their dietary intake data alone.
  Other Names: Dietary intake Group
  Arms: Level 1
Behavioral: Level 2 — Level or Group 2: Participants will receive personalised dietary advice taking dietary intake and phenotypic data into account.
  Other Names: Dietary Intake + Phenotype Group
  Arms: Level 2
Behavioral: Level 3 — Level or group 3: Participants will receive personalised dietary advice taking dietary intake, phenotypic and genotypic data into account.
  Other Names: Dietary + Phenotype + Genotype Group
  Arms: Level 3
Behavioral: Level 0 — Level 0 - Control group - Investigators will provide non-personalized dietary advice for improved food choice based on standard population healthy eating guidelines.
  Other Names: Control group
  Arms: Level 0

SUMMARY:
The concept of personalised nutrition emerged following the sequencing of the human genome in 2000. It was hoped that with the identification of gene nutrient interactions, an individual's response and susceptibility to particular diets would be better understood and therefore appropriate dietary modifications could be made to optimise health and lower disease risk. Then Food4Me aims to study the development of personalized nutrition at three levels and determine whether providing more personalised dietary advice leads to better compliance and health outcomes compared to standard population advice.

The hypotheses to be tested in the Food4Me study are as follows:

* Personalisation of dietary advice assists and/or motivates consumers to eat a healthier diet and follow a healthier lifestyle (in comparison with "impersonal" [conventional] dietary advice).
* Personalisation based on individualised biochemical (phenotypic) and/or genetic information is more effective in assisting and/or motivating study participants to make, and to sustain, appropriate healthy changes to their usual (habitual) diet and lifestyle.

DETAILED DESCRIPTION:
To achieve the Food4me aims, investigators will undertake a large multi-centre proof-of-principle study carried out across 7 EU countries on options for the delivery of personalised nutrition.

Recruitment Centres

Recruitment to the Food4Me intervention study will be carried out using identical protocols in 7 centres across the EU involving a total of 1,288 study participants i.e. 184 participants per country. The Proof-of-Proof of Principle study centres involve in the recruitment are:

* University College Dublin, Ireland.
* University of Maastricht, Netherlands.
* Universidad de Navarra, Spain.
* Harokopio University, Greece.
* The University of Reading, Uk
* National Food and Nutrition Institute, Poland.
* Technische Universitaet Muenchen, German.

Study design

Then, each proof-of-principle centre will recruit a sample of 184 participants and with 46 subjects will be randomly assigned each of the following levels of personalised nutrition:

* Level 0: Control group - will receive non-personalized dietary advice for improved food choice based on standard population healthy eating guidelines.
* Level 1: Personalised dietary advice based on dietary intake data alone.
* Level 2: Personalised dietary advice taking dietary intake and phenotypic data into account.
* Level 3: Personalised dietary advice taking dietary intake, phenotypic and genotypic data into account.

The study has been designed to mimic a fully Internet delivered personalized nutrition service. The route to recruitment will be via the Internet to mimic the real life conditions for a "proof-of-principle" study. However, to ensure adequate recruitment to this scientific study, the recruitment of study participants will be also based on local and national advertising of the service through internet, radio advertisements, other advertisements, use of social media or face to face meetings.

Only participants aged 18 years of age and above will be included in the study. A minimal set of exclusion criteria will be applied (subject under 18 years old, pregnant or lactating, no or limited access to internet, following a prescribed diet for any reason, including weight loss in the last 3 months, Insulin dependent diabetes, celiac disease, Crohn's, or any metabolic disease or condition that alters nutritional requirements, such as diabetes. Other than balancing the male to female ratio among recruits (with not more than a 70/30 or 30/70 distribution of males and females in each group) and balancing the age ratio (with not more than a 70/30 or 30/70 distribution of participants <45 years and > 45 years old in each group) no other stratification will be applied since the objective is to complete the proof-of-principle study in as real setting as possible. All age and sex stratification will be applied before randomisation of the participants to each level / group of personalised nutrition (0, 1, 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years old

Exclusion Criteria:

* Subject under 18 years old.
* Pregnant or lactating.
* No or limited access to internet.
* Following a prescribed diet for any reason, including weight loss in the last 3 months.
* Subjects under medication for Insulin dependent diabetes, celiac disease, Crohn's or any metabolic disease or condition that alters nutritional requirements, such as diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1607 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Dietary Intake at 3 and 6 months | Baseline, month 3 and 6.
  Habitual (usual) dietary intake will be measured using an on-line Food Frequency Questionnaire (FFQ). Intakes of nutrients will be computed using a food composition data base which has been augmented with country-specific food composition data. Changes in dietary pattern will be compared between baseline and month 3 and 6 in all participants.

SECONDARY OUTCOMES:
Change from baseline in phenotypic and Metabolic biomarkers at 3 and 6 month | baseline, month 3 and 6
  Obesity-related phenotypes (Weight [kg], BMI [kg/m^2], waits circumference [cm]Changes in glucose [mg/dl]),and metabolic-related markers (glucose [mg/dl], fatty acid [%]and total cholesterol [mg/dl]), will be measured at baseline, month 3 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: John Mathers, Professor, Principal Investigator — Newcastle University, United Kingdom; Mike Gibney, Professor, Study Director — University College Dublin, Ireland; Wim Saris, Professor, Principal Investigator — •Universiteit Maastricht, Netehrlands; Alfredo Martinez, Professor, Principal Investigator — University of Navarra, Spain; Julie Lovegrove, Professor, Principal Investigator — University of Reading, United Kingdom; Yannis Manios, Professor, Principal Investigator — Harokopio University, Athens, Greece; Iwona Traczyk, Professor, Principal Investigator — National Food and Nutrition Institute, Warsaw, Poland; Hannelore Daniel, Professor, Principal Investigator — Technische Universitaet Muenchen, Germany
Locations (8):
- Technische Universitaet Muenchen, München, Germany
- The Harokopio University, Athens, Greece
- University College Dublin, Dublin, Ireland
- Maastricht University, Maastricht, Netherlands
- National Food and Nutritional Institute, Warsaw, Poland
- University of Navarra, Navarra, Spain
- United Kingdom (2):
  - Newcastle University, Newcastle
  - University of Reading, Reading

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request from the Project leader Professor Mike Gibney and Professor John Mathers.

REFERENCES:
- [Derived] Livingstone KM, Brayner B, Celis-Morales C, Moschonis G, Manios Y, Traczyk I, Drevon CA, Daniel H, Saris WHM, Lovegrove JA, Gibney M, Gibney ER, Brennan L, Martinez JA, Mathers JC. Associations between dietary patterns, FTO genotype and obesity in adults from seven European countries. Eur J Nutr. 2022 Sep;61(6):2953-2965. doi: 10.1007/s00394-022-02858-3. Epub 2022 Mar 21. PMID 35307761
- [Derived] Livingstone KM, Celis-Morales C, Navas-Carretero S, San-Cristobal R, Forster H, Woolhead C, O'Donovan CB, Moschonis G, Manios Y, Traczyk I, Gundersen TE, Drevon CA, Marsaux CFM, Fallaize R, Macready AL, Daniel H, Saris WHM, Lovegrove JA, Gibney M, Gibney ER, Walsh M, Brennan L, Martinez JA, Mathers JC; Food4Me Study. Personalised nutrition advice reduces intake of discretionary foods and beverages: findings from the Food4Me randomised controlled trial. Int J Behav Nutr Phys Act. 2021 Jun 7;18(1):70. doi: 10.1186/s12966-021-01136-5. PMID 34092234
- [Derived] Celis-Morales C, Livingstone KM, Petermann-Rocha F, Navas-Carretero S, San-Cristobal R, O'Donovan CB, Moschonis G, Manios Y, Traczyk I, Drevon CA, Daniel H, Marsaux CFM, Saris WHM, Fallaize R, Macready AL, Lovegrove JA, Gibney M, Gibney ER, Walsh M, Brennan L, Martinez JA, Mathers JC; Food4Me Study. Frequent Nutritional Feedback, Personalized Advice, and Behavioral Changes: Findings from the European Food4Me Internet-Based RCT. Am J Prev Med. 2019 Aug;57(2):209-219. doi: 10.1016/j.amepre.2019.03.024. Epub 2019 Jun 25. PMID 31248745
- [Derived] Macready AL, Fallaize R, Butler LT, Ellis JA, Kuznesof S, Frewer LJ, Celis-Morales C, Livingstone KM, Araujo-Soares V, Fischer AR, Stewart-Knox BJ, Mathers JC, Lovegrove JA. Application of Behavior Change Techniques in a Personalized Nutrition Electronic Health Intervention Study: Protocol for the Web-Based Food4Me Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 9;7(4):e87. doi: 10.2196/resprot.8703. PMID 29631993
- [Derived] San-Cristobal R, Navas-Carretero S, Celis-Morales C, Livingstone KM, Stewart-Knox B, Rankin A, Macready AL, Fallaize R, O'Donovan CB, Forster H, Woolhead C, Walsh MC, Lambrinou CP, Moschonis G, Manios Y, Jarosz M, Daniel H, Gibney ER, Brennan L, Gundersen TE, Drevon CA, Gibney M, Marsaux CFM, Saris WHM, Lovegrove JA, Frewer LJ, Mathers JC, Martinez JA; Food4Me Study. Capturing health and eating status through a nutritional perception screening questionnaire (NPSQ9) in a randomised internet-based personalised nutrition intervention: the Food4Me study. Int J Behav Nutr Phys Act. 2017 Dec 11;14(1):168. doi: 10.1186/s12966-017-0624-6. PMID 29228998
- [Derived] Celis-Morales C, Marsaux CF, Livingstone KM, Navas-Carretero S, San-Cristobal R, Fallaize R, Macready AL, O'Donovan C, Woolhead C, Forster H, Kolossa S, Daniel H, Moschonis G, Mavrogianni C, Manios Y, Surwillo A, Traczyk I, Drevon CA, Grimaldi K, Bouwman J, Gibney MJ, Walsh MC, Gibney ER, Brennan L, Lovegrove JA, Martinez JA, Saris WH, Mathers JC. Can genetic-based advice help you lose weight? Findings from the Food4Me European randomized controlled trial. Am J Clin Nutr. 2017 May;105(5):1204-1213. doi: 10.3945/ajcn.116.145680. Epub 2017 Apr 5. PMID 28381478
- [Derived] O'Donovan CB, Walsh MC, Forster H, Woolhead C, Celis-Morales C, Fallaize R, Macready AL, Marsaux CF, Navas-Carretero S, San-Cristobal R, Kolossa S, Mavrogianni C, Lambrinou CP, Moschonis G, Godlewska M, Surwillo A, Bouwman J, Grimaldi K, Traczyk I, Drevon CA, Daniel H, Manios Y, Martinez JA, Saris WH, Lovegrove JA, Mathers JC, Gibney MJ, Brennan L, Gibney ER. The impact of MTHFR 677C --> T risk knowledge on changes in folate intake: findings from the Food4Me study. Genes Nutr. 2016 Sep 29;11:25. doi: 10.1186/s12263-016-0539-x. eCollection 2016. PMID 27708721
- [Derived] Livingstone KM, Celis-Morales C, Hoeller U, Lambrinou CP, Moschonis G, Macready AL, Fallaize R, Baur M, Roos FF, Bendik I, Grimaldi K, Navas-Carretero S, San-Cristobal R, Weber P, Drevon CA, Manios Y, Traczyk I, Gibney ER, Lovegrove JA, Saris WH, Daniel H, Gibney M, Martinez JA, Brennan L, Hill TR, Mathers JC; Food4Me Study. Weekday sunlight exposure, but not vitamin D intake, influences the association between vitamin D receptor genotype and circulating concentration 25-hydroxyvitamin D in a pan-European population: the Food4Me study. Mol Nutr Food Res. 2017 Feb;61(2). doi: 10.1002/mnfr.201600476. Epub 2016 Nov 11. PMID 27682437
- [Derived] Fallaize R, Celis-Morales C, Macready AL, Marsaux CF, Forster H, O'Donovan C, Woolhead C, San-Cristobal R, Kolossa S, Hallmann J, Mavrogianni C, Surwillo A, Livingstone KM, Moschonis G, Navas-Carretero S, Walsh MC, Gibney ER, Brennan L, Bouwman J, Grimaldi K, Manios Y, Traczyk I, Drevon CA, Martinez JA, Daniel H, Saris WH, Gibney MJ, Mathers JC, Lovegrove JA; Food4Me Study. The effect of the apolipoprotein E genotype on response to personalized dietary advice intervention: findings from the Food4Me randomized controlled trial. Am J Clin Nutr. 2016 Sep;104(3):827-36. doi: 10.3945/ajcn.116.135012. Epub 2016 Aug 10. PMID 27510539
- [Derived] Livingstone KM, Celis-Morales C, Lara J, Woolhead C, O'Donovan CB, Forster H, Marsaux CF, Macready AL, Fallaize R, Navas-Carretero S, San-Cristobal R, Kolossa S, Tsirigoti L, Lambrinou CP, Moschonis G, Surwillo A, Drevon CA, Manios Y, Traczyk I, Gibney ER, Brennan L, Walsh MC, Lovegrove JA, Martinez JA, Saris WH, Daniel H, Gibney M, Mathers JC. Clustering of adherence to personalised dietary recommendations and changes in healthy eating index within the Food4Me study. Public Health Nutr. 2016 Dec;19(18):3296-3305. doi: 10.1017/S1368980016001932. Epub 2016 Aug 8. PMID 27499187
- [Derived] Livingstone KM, Celis-Morales C, Macready AL, Fallaize R, Forster H, Woolhead C, O'Donovan CB, Marsaux CF, Navas-Carretero S, San-Cristobal R, Kolossa S, Tsirigoti L, Lambrinou CP, Moschonis G, Surwillo A, Drevon CA, Manios Y, Traczyk I, Gibney ER, Brennan L, Walsh MC, Lovegrove JA, Martinez JA, Saris WH, Daniel H, Gibney M, Mathers JC. Characteristics of European adults who dropped out from the Food4Me Internet-based personalised nutrition intervention. Public Health Nutr. 2017 Jan;20(1):53-63. doi: 10.1017/S1368980016002020. Epub 2016 Aug 5. PMID 27492149
- [Derived] Forster H, Walsh MC, O'Donovan CB, Woolhead C, McGirr C, Daly EJ, O'Riordan R, Celis-Morales C, Fallaize R, Macready AL, Marsaux CF, Navas-Carretero S, San-Cristobal R, Kolossa S, Hartwig K, Mavrogianni C, Tsirigoti L, Lambrinou CP, Godlewska M, Surwillo A, Gjelstad IM, Drevon CA, Manios Y, Traczyk I, Martinez JA, Saris WH, Daniel H, Lovegrove JA, Mathers JC, Gibney MJ, Gibney ER, Brennan L. A Dietary Feedback System for the Delivery of Consistent Personalized Dietary Advice in the Web-Based Multicenter Food4Me Study. J Med Internet Res. 2016 Jun 30;18(6):e150. doi: 10.2196/jmir.5620. PMID 27363307
- [Derived] Livingstone KM, Celis-Morales C, Navas-Carretero S, San-Cristobal R, Macready AL, Fallaize R, Forster H, Woolhead C, O'Donovan CB, Marsaux CF, Kolossa S, Tsirigoti L, Lambrinou CP, Moschonis G, Godlewska M, Surwillo A, Drevon CA, Manios Y, Traczyk I, Gibney ER, Brennan L, Walsh MC, Lovegrove JA, Saris WH, Daniel H, Gibney M, Martinez JA, Mathers JC; Food4Me Study. Effect of an Internet-based, personalized nutrition randomized trial on dietary changes associated with the Mediterranean diet: the Food4Me Study. Am J Clin Nutr. 2016 Aug;104(2):288-97. doi: 10.3945/ajcn.115.129049. Epub 2016 Jun 29. PMID 27357094
- [Derived] Marshall SJ, Livingstone KM, Celis-Morales C, Forster H, Fallaize R, O'Donovan CB, Woolhead C, Marsaux CF, Macready AL, Navas-Carretero S, San-Cristobal R, Kolossa S, Tsirigoti L, Lambrinou CP, Moschonis G, Godlewska M, Surwillo A, Drevon CA, Manios Y, Traczyk I, Martinez JA, Saris WH, Daniel H, Gibney ER, Brennan L, Walsh MC, Lovegrove JA, Gibney M, Mathers JC; Food4Me Study. Reproducibility of the Online Food4Me Food-Frequency Questionnaire for Estimating Dietary Intakes across Europe. J Nutr. 2016 May;146(5):1068-75. doi: 10.3945/jn.115.225078. Epub 2016 Apr 6. PMID 27052541
- [Derived] Marsaux CF, Celis-Morales C, Livingstone KM, Fallaize R, Kolossa S, Hallmann J, San-Cristobal R, Navas-Carretero S, O'Donovan CB, Woolhead C, Forster H, Moschonis G, Lambrinou CP, Surwillo A, Godlewska M, Hoonhout J, Goris A, Macready AL, Walsh MC, Gibney ER, Brennan L, Manios Y, Traczyk I, Drevon CA, Lovegrove JA, Martinez JA, Daniel H, Gibney MJ, Mathers JC, Saris WH. Changes in Physical Activity Following a Genetic-Based Internet-Delivered Personalized Intervention: Randomized Controlled Trial (Food4Me). J Med Internet Res. 2016 Feb 5;18(2):e30. doi: 10.2196/jmir.5198. PMID 26851191
- [Derived] Marsaux CF, Celis-Morales C, Fallaize R, Macready AL, Kolossa S, Woolhead C, O'Donovan CB, Forster H, Navas-Carretero S, San-Cristobal R, Lambrinou CP, Moschonis G, Surwillo A, Godlewska M, Goris A, Hoonhout J, Drevon CA, Manios Y, Traczyk I, Walsh MC, Gibney ER, Brennan L, Martinez JA, Lovegrove JA, Gibney MJ, Daniel H, Mathers JC, Saris WH. Effects of a Web-Based Personalized Intervention on Physical Activity in European Adults: A Randomized Controlled Trial. J Med Internet Res. 2015 Oct 14;17(10):e231. doi: 10.2196/jmir.4660. PMID 26467573
- [Derived] Hallmann J, Kolossa S, Gedrich K, Celis-Morales C, Forster H, O'Donovan CB, Woolhead C, Macready AL, Fallaize R, Marsaux CF, Lambrinou CP, Mavrogianni C, Moschonis G, Navas-Carretero S, San-Cristobal R, Godlewska M, Surwillo A, Mathers JC, Gibney ER, Brennan L, Walsh MC, Lovegrove JA, Saris WH, Manios Y, Martinez JA, Traczyk I, Gibney MJ, Daniel H; Food4Me Study. Predicting fatty acid profiles in blood based on food intake and the FADS1 rs174546 SNP. Mol Nutr Food Res. 2015 Dec;59(12):2565-73. doi: 10.1002/mnfr.201500414. Epub 2015 Sep 30. PMID 26346302
- [Derived] Celis-Morales C, Livingstone KM, Woolhead C, Forster H, O'Donovan CB, Macready AL, Fallaize R, Marsaux CFM, Tsirigoti L, Efstathopoulou E, Moschonis G, Navas-Carretero S, San-Cristobal R, Kolossa S, Klein UL, Hallmann J, Godlewska M, Surwillo A, Drevon CA, Bouwman J, Grimaldi K, Parnell LD, Manios Y, Traczyk I, Gibney ER, Brennan L, Walsh MC, Lovegrove JA, Martinez JA, Daniel H, Saris WHM, Gibney M, Mathers JC. How reliable is internet-based self-reported identity, socio-demographic and obesity measures in European adults? Genes Nutr. 2015 Sep;10(5):28. doi: 10.1007/s12263-015-0476-0. Epub 2015 Jul 5. PMID 26143178
- See also: Study Official webpage — http://food4me.org/